CLINICAL TRIAL: NCT05605470
Title: A Phase 2 Study to Evaluate the Immunogenicity and Safety of ChulaCov19 BNA159 and ChulaCov19 BNA159.2 Vaccines as a Booster Dose in Adults Who Have Received a Previous Booster Dose of an Authorized/Approved COVID-19 Vaccine
Brief Title: Immunogenicity and Safety of ChulaCov19 BNA159 and ChulaCov19 BNA159.2 Vaccines as a Booster Dose in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technovalia, Pty Ltd (Industry)
Collaborators: Chulalongkorn University (Other); BioNet-Asia (Unknown); Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TVL-ChulaVac005
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: COVID-19, SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A: Arm 1 (1 dose of ChulaCov19 BNA159 vaccine) (Experimental): Participants will be randomized to receive ChulaCov19 BNA159 vaccine (50 mcg) given by IM (n=55)
  Interventions: Biological: ChulaCov19 BNA159 vaccine (50 mcg)
- Part A: Arm 2 (one dose of active comparator vaccine) (Active Comparator): Participants will be randomized to receive Comirnaty® (Pfizer/BNT) vaccine (30 mcg) given by IM (n=25)
  Interventions: Biological: Pfizer/BNT vaccine (30 mcg)
- Part B: Arm 3 (one dose of COMVIGEN vaccine) (Experimental): Participants will be randomized to receive ChulaCov19 BNA159.2 (COMVIGEN) vaccine (50 mcg) given by IM (n=70)
  Interventions: Biological: COMVIGEN (ChulaCov19 BNA159.2) vaccine (50 mcg)

INTERVENTIONS:
Biological: ChulaCov19 BNA159 vaccine (50 mcg) — Single dose of ChulaCov19 BNA159 vaccine 0.5 ml will be given by IM at Day 1
  Arms: Part A: Arm 1 (1 dose of ChulaCov19 BNA159 vaccine)
Biological: Pfizer/BNT vaccine (30 mcg) — Single dose of Pfizer/BNT vaccine 0.3 ml will be given by IM at Day 1
  Arms: Part A: Arm 2 (one dose of active comparator vaccine)
Biological: COMVIGEN (ChulaCov19 BNA159.2) vaccine (50 mcg) — Single dose of COMVIGEN vaccine 0.5 ml will be given by IM at Day 1
  Arms: Part B: Arm 3 (one dose of COMVIGEN vaccine)

SUMMARY:
This clinical trial is designed to assess the safety, tolerability and immunogenicity of a single dose of ChulaCov19 BNA159 and ChulaCov19 BNA159.2 vaccines as a booster dose, given at least 3 months after receipt of a previous booster dose of any authorized/approved COVID-19 vaccine.

DETAILED DESCRIPTION:
This is a phase II, randomised open-label trial in which 150 healthy males and non-pregnant females aged 18-64 years, will be recruited from multi-sites in Australia. This is a 2-part study (Part A and Part B). In Part A, the randomisation will be a 2:1 design to receive either ChulaCov19 BNA159 vaccine or Comirnaty Pfizer/BNT vaccine. In Part B, participants will receive only ChulaCov19 BNA159.2 (Bivalent, COMVIGEN) vaccine. Participants in part A and B will be followed up using a combination of an-site and telephone visits for assessment of safety and immunogenicity for 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male or female aged 18 - 64 (inclusive) at the time of enrolment
2. Must have completed a primary course of 2 doses of any approved COVID-19 vaccine and 3 months or more have passed since receipt of last booster dose (1 or 2 prior booster doses for a total of 3 or 4 doses) as described in Table 1
3. Must be able to communicate effectively with study personnel and considered reliable, willing, and cooperative in terms of compliance with the protocol requirements
4. Participants must sign the written informed consent form prior to undertaking any protocol-related procedures
5. SARS-CoV-2 rapid antigen test is negative at Day 1 (the day of receiving the study booster dose)
6. Does not intend to receive any other authorized/approved COVID-19 vaccine at the time of enrolment and up to 3 months of the study
7. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), practice true abstinence or, if engaged in sexual relations with a female of childbearing potential, the participants and their partner must use an acceptable, highly effective, dual contraceptive method* from Screening and for a period of at least 90 days after vaccination
8. A female participant is eligible if she is not pregnant, or breastfeeding indicated by one of the following conditions:

   1. With childbearing potential: she agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the study intervention administration until at least 90 days after the study intervention administration, or
   2. With non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile. If the participant is < 1 year post-menopausal, an FSH test may be conducted to establish childbearing potential.
9. Participants must be in general good health* based on medical history and physical examination, as determined by the PI at Screening.
10. Participants must agree to refrain from donating blood, plasma, ova, sperm, or organs during the whole study.

Exclusion Criteria:

1. History of a systemic hypersensitivity or life-threatening reaction to a vaccine containing any of the same or similar substances.
2. History of test-confirmed by PCR or rapid antigen test to SARS-CoV-2 COVID-19 infection within 3 months prior to randomisation.
3. Presence of clinically significant medical history*, unstable chronic or acute disease that, in the opinion of the PI, may increase the risk of exposure to the investigational vaccine
4. History of having any significant side effects after receipt of any other COVID-19 vaccine eg. endocarditis, pericarditis or myocarditis. History of any severe reactogenic side effects or other medical illness that were thought to be associated with vaccine.
5. Presence of an acute illness* or with fever at 38.00 C or more within 72 hours prior to vaccination.
6. Bleeding disorders or taking an anticoagulant or anti-platelet agent that may contraindicate for intramuscular injection based on Investigator's judgment
7. Inadequate venous access to allow the collection of blood samples.
8. Received any prophylactic or therapeutic vaccine, biologic product, device or blood product, within 4 weeks of vaccination or 5 half-lives (whichever is longer) or anticipate doing so in the follow-up period defined for this study. For influenza vaccine, however, can be administered up to 14 days prior to randomization and following Visit 3 (Day 29+3) blood sample collection.
9. History of ever had an anaphylaxis reaction to food, medication, or vaccination.
10. Participant is immunosuppressed as caused by disease or immunosuppressive therapy or anticipated need to use of any chemotherapy or immunosuppressive agents* within the next 6 months.
11. Participation in any of the other investigational trials of vaccines, therapeutic, or medical devices 12 weeks before or during the 6 months of this study.
12. Received immunoglobulins and/or any blood or blood products within 3 months before vaccination day or plans to receive any blood or blood products at any time during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Numbers and percentage of participants with immediate adverse events | within 30 minutes post vaccination
  Numbers and percentage of participants who have had immediate post-immunization reactions within 30 minutes post- vaccination
Part A and Part B: Numbers and percentage of participants with solicited local or systemic reactions | within 7-day post-vaccination
  Numbers and percentage of participants who have had solicited local or systemic reactions within 7-day post-vaccination
Part A and Part B: Numbers and percentage of participants with adverse events (AEs) | 28-day post-vaccination
  Numbers and percentage of participants who have had adverse events (AEs) within 28-day post-vaccination
Part A and Part B:Numbers and percentage of participants with serious adverse events (SAEs), medically attended adverse events (MAAEs) and New Onset Chronic Medical Condition (NOCMCs) | 6 months post-vaccination
  Numbers and percentage of participants who have had SAEs, MAAEs, NOCMCs within 6 months post-vaccination
Geometric mean titres (GMTs) of SARS-CoV-2-specific serum neutralising antibody as measured by psVNT-50 against wild type and/or Omicron BA.4/BA.5 | Baseline, 28-day post-vaccination
  GMTs and their 95%CI of SARS-CoV-2-specific serum neutralising antibody as measured by psVNT-50 against wild type (Part A and B) and/or Omicron BA.4/BA.5 (Part B) will be reported at baseline (before vaccination) and 28 days post-vaccination.
Geometric mean fold rises (GMFRs) of SARS-CoV-2-specific serum neutralising titres as measured by psVNT-50 against wild type and/or Omicron BA.4/BA.5 | Baseline, 28-day post-vaccination
  GMFRs and their 95%CI of SARS-CoV-2-specific serum neutralising titres as measured by psVNT-50 against wild type (Part A and B) and/or Omicron BA.4/BA.5 (Part B) will be reported from baseline to 28 days post-vaccination.
Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by psVNT-50 against wild type and/or Omicron BA.4/BA.5 | 28 days post-vaccination.
  Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by psVNT-50 against wild type (Part A and B) and/or Omicron BA.4/BA.5 (Part B) will be reported at 28 days post-vaccination.

SECONDARY OUTCOMES:
GMTs of SARS-CoV-2-specific serum neutralising antibody as measured by psVNT-50 against Omicron BA.4/BA.5 and/or other clinically relevant variants of concerns (VOCs) | Baseline, 28-day post-vaccination
  GMTs and their 95%CI of SARS-CoV-2-specific serum neutralising antibody as measured by psVNT-50 against Omicron BA.4/BA.5 (Part A) and/or other clinically relevant VOCs (Part A and B) will be reported at baseline (before vaccination) and 28 days post-vaccination.
GMFRs of SARS-CoV-2-specific serum neutralising titres as measured by psVNT-50 against Omicron BA.4/BA.5 and/or other clinically relevant VOCs | Baseline, 28-day post-vaccination
  GMFR and their 95%CI of SARS-CoV-2-specific serum neutralising titres as measured by psVNT-50 against Omicron BA.4/BA.5 (Part A) and/or other clinically relevant VOCs (Part A and B) will be reported from baseline to 28 days post-vaccination.
Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by psVNT-50 against Omicron BA.4/BA.5 and/or other clinically relevant VOCs | 28-day post-vaccination
  Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by psVNT-50 against Omicron BA.4/BA.5 (Part A) and/or other clinically relevant VOCs (Part A and B) will be reported at 28 days post-vaccination.
GMTs of SARS-CoV-2-specific serum neutralising antibody as measured by MicroVNT-50 against wild type | Baseline, 28-day post-vaccination
  Part A and Part B: GMTs and their 95%CI of SARS-CoV-2-specific serum neutralising antibody as measured by MicroVNT-50 against wild type will be reported at baseline (before vaccination) and 28 days post-vaccination.
GMFRs of SARS-CoV-2-specific serum neutralising titres as measured by MicroVNT-50 against wild type | Baseline to 28 days post-vaccination.
  Part A and Part B: GMFR and their 95%CI of SARS-CoV-2-specific serum neutralising titres as measured by MicroVNT-50 against wild type will be reported from baseline to 28 days post-vaccination.
Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by MicroVNT-50 against wild type | 28 days post-vaccination
  Part A and Part B: Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV-2-specific serum neutralising antibody titres as measured by MicroVNT-50 against wild type will be reported at 28 days post-vaccination.
GMTs of SARS-CoV2-RBD-binding (anti-RBD) and Spike-binding (anti-S) IgG antibodies as measured by ELISA against wild type and Omicron. | Baseline and 28 days post-vaccination.
  GMTs and their 95%CI of anti-RBD and anti-S IgG antibodies as measured by ELISA against wild type (Part A and B) and Omicron (Part B) will be reported at baseline (before vaccination) and 28 days post-vaccination.
GMFRs of SARS-CoV2-RBD-binding (anti-RBD) and Spike-binding (anti-S) IgG antibodies as measured by ELISA against wild type and Omicron. | Baseline to 28 days post-vaccination.
  GMFR and their 95%CI of anti-RBD and anti-S IgG antibodies as measured by ELISA against wild type (Part A and B) and Omicron (Part B) will be reported from baseline to 28 days post-vaccination.
Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of SARS-CoV2-RBD-binding (anti-RBD) and Spike-binding (anti-S) IgG antibodies as measured by ELISA against wild type and Omicron. | 28 days post-vaccination
  Percentage of participants who achieved a greater than or equal to 4-fold rise from before vaccination of anti-RBD and anti-S IgG antibodies as measured by ELISA against wild type (Part A and B) and Omicron (Part B) will be reported at 28 days post-vaccination
Geometric mean (GM) and/or median number of SARS-CoV2-specific T-cell responses (spot-forming cells (SFC) per 1 million PBMCs) measured by IFNγ-ELISpot assay against wild-type peptides | Baseline and 28 days post-vaccination.
  Part A and Part B: GM and/or median number of SFC per 1 million PBMCs measured by IFNγ-ELISpot assay against wild-type peptides will be reported at baseline (before vaccination) and 28 days post-vaccination
GMFRs of number of SFC per 1 million PBMCs measured by IFNγ-ELISpot assay against wild-type peptides | Baseline to 28 days post-vaccination.
  Part A and Part B: GMFR and their 95%CI of number of SFC per 1 million PBMCs measured by IFNγ-ELISpot assay against wild-type peptides will be reported from baseline to 28 days post-vaccination.
GM and/or median number of % Spike specific CD4 and CD8 T-cells as measured by Intracellular Cytokine Staining (ICS) assay | Baseline and 28 days post-vaccination
  Part A and Part B: GM and/or median number of % Spike specific CD4 and CD8 T-cells as measured by ICS assay (from the first 25 subjects from the ChulaCov19 group, the comparator group and COMVIGEN) will be reported at baseline (before vaccination) and 28 days post-vaccination.
GMFR of % Spike-specific CD4 and CD8 T-cells as measured by ICS assay | Baseline to 28 days post-vaccination.
  Part A and Part B: GMFR of % Spike-specific CD4 and CD8 T-cells as measured by ICS assay (from the first 25 subjects from the ChulaCov19 group, the comparator group and COMVIGEN) will be reported from baseline to 28 days post-vaccination.
GM and/or median number of Th1/Th2 ratio as measured by ICS assay | Baseline and 28 days post-vaccination
  Part A and Part B: GM and/or median number of Th1/Th2 ratio as measured by ICS assay (from the first 25 subjects from the ChulaCov19 group, the comparator group and COMVIGEN) will be reported at baseline (before vaccination) and 28 days post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrunghtam, MD, Study Director — Chulalongkorn University
Locations (5):
- Australia (5):
  - Paratus research Canberra Clinic, Bruce, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - The Children's Hospital at Westmead Sydney, Westmead, New South Wales
  - Paratus Clinical Research- Brisbane Clinic, Albion, Queensland

IPD SHARING:
Plan to Share IPD: No